CLINICAL TRIAL: NCT06802263
Title: Assessing Accuracy and Precision of Home Quantitative Urine Beta hCG With Serum for Pregnancy of Unknown Location (CONNECT)
Brief Title: MIRA CONNECT Study
Acronym: CONNECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-1954
Record Dates: First submitted 2025-01-06; First posted 2025-01-31 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy of Unknown Location (PUL)
Keywords: pregnancy; unknown location; b-hCG

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- CNTRL: Non-pregnant control patients (Sham Comparator): Non-pregnant patients will use the pregnancy test device
  Interventions: Diagnostic Test: at-home quantitative urine b-hCG test
- PUL: Pregnancy unknown location diagnosis (Active Comparator): Pregnant patients with unknown location diagnosis will use the pregnancy test device
  Interventions: Diagnostic Test: at-home quantitative urine b-hCG test

INTERVENTIONS:
Diagnostic Test: at-home quantitative urine b-hCG test — Cases will begin performing urine and serum hCG testing 24 hours after the initial hCG level. Urine hCG testing will be performed on the first morning urine at home and participants will limit water for at least 8 hours before testing. Serum hCG testing will occur at a UCHealth laboratory before 10 am and within 2 hours of the urine test to allow for the comparison of the values. Both urine and serum hCG testing will then occur daily x 7 days, or until a medical or surgical intervention is indicated. If serum testing is indicated on a weekend, patients will present to the UCH Infusion Center.
  Non-pregnant controls will test the first morning urine at home and undergo serum hCG testing in a UCHealth lab on the 4th and 6th day of the menstrual cycle. All urine hCG values will be recorded in the Mira home kit and evaluated in comparison to serum hCG levels.

SUMMARY:
The goal of this pilot study is to assess the accuracy and precision of an at-home quantitative urine beta hCG (b-hCG) test in the management of pregnancy of unknown location (PUL).

DETAILED DESCRIPTION:
This study proposes to test the ability of the Mira urine hCG testing kit to accurately and precisely quantify urine beta hCG testing in women with PUL, thus preventing unnecessary travel time to medical care, time lost from work, costs of childcare services, anxiety, and lack of adherence to medical recommendations.

Aim 1: Assess the accuracy and precision of an at-home quantitative urine b-hCG test in the management of pregnancy of unknown location (PUL). Hypothesis: The Mira quantitative home urine pregnancy test will accurately and precisely quantify beta hCG levels in patients with PUL.

Approach: The study team will recruit 30 women with a diagnosed pregnancy of unknown location (cases) and non-pregnant 5 controls. Potential participants may be identified in the emergency department (ED), inpatient floor, or University of Colorado Health (UC Health) or School of Medicine (CU Medicine) outpatient clinics. Once a diagnosis of PUL is established, cases will be provided with a Mira home testing device.

Cases will begin performing urine and serum hCG testing 24 hours after the initial hCG level. Urine hCG testing will be performed on the first morning urine at home and participants will limit water for at least 8 hours before testing. Serum hCG testing will occur at a UCHealth laboratory before 10 am and within 2 hours of the urine test to allow for the comparison of the values. Both urine and serum hCG testing will then occur daily x 7 days, or until a medical or surgical intervention is indicated. If serum testing is indicated on a weekend, patients will present to the UCH Infusion Center.

Non-pregnant controls will test the first morning urine at home and undergo serum hCG testing in a UCHealth lab on the 4th and 6th day of the menstrual cycle. All urine hCG values will be recorded in the Mira home kit and evaluated in comparison to serum hCG levels.

Aim 2: Assess patient satisfaction with the Mira at-home quantitative urine b-hCG test in the management of PUL. Hypothesis: Participants will find the Mira at-home quantitative urine beta hCG test easy to use and will be satisfied with communication with the provider team.

Approach: Participants will complete a survey at the end of the study to assess ease of use and satisfaction with at-home testing as a method of management for PUL.

Research Methods

As part of this pilot study, the investigator aims to enroll a cohort of 30 female patients with a diagnosis of PUL. Participants will perform the urine pregnancy testing at home and undergo the quantitative serum b-hCG testing at UCH. The investigator will also perform testing on five non-pregnant female control subjects in the same age group. Enrolled participants will have eight study visits with the following data collected: Urine b-hCG and serum b-hCG

A. Study Design and Research Methods: This will be a pilot study. Patients with pregnancy of unknown location may be recruited in the OBGYN ambulatory clinics or in the Emergency Department. Non-pregnant control subjects will be recruited from the UCH AOP OBGYN ambulatory clinics. The PI does have a clinical relationship with both of these patient populations.

The research coordinator will identify patients who meet study criteria and contact the patient to explain the study and obtain consent/assent, if interested. The study visits for the serum b-hCG levels will be scheduled at that time. Study visits for cases will occur daily for 7 days after the PUL has been established. Non-pregnant controls will undergo home urine testing and serum HCG testing on the 4th and 6th day of their menstrual cycle. Day 1 of their menstrual cycle is defined as the first day of flow that soaks more than one panty liner. On days 4 and 6 of their cycle, control participants will test their first morning urine at home and undergo serum hCG testing in a UCHealth lab before 10am.

The Principal Investigator has worked with the Mira team to develop a process so that Mira does not receive any identifying information about the study participants as well as a way to blind the participants to their results.

All study participants will be required to download the Mira Fertility & Cycle Tracking app onto their smartphone. This app is supported on both iOS and Android smartphones. Participants will login to the system with unique credentials provided by Mira with a study ID attached (e.g. Mira001, Mira002 and so on). The quantitative hCG will be visible on the device screen as Mira does not have a way to blind this data. However, participants will be taught that these numbers should not be used to inform clinical care.

The Mira device connects to the app via Bluetooth and all data will be transferred to a web-based cloud supported by Amazon Web Services (AWS). Mira will send the data to the study team, which will then be entered into the study REDCap database. Data within the app are not available to the patient nor their clinical team.

All participants:

The first study visit will occur at the time of diagnosis and includes:

* Past medical history, gynecologic and obstetric history obtained via REDCap questionnaire by the study coordinator at time of study enrollment
* Download of Mira Fertility and Cycle Tracker app
* Login to the app using generic credentials provided by Mira.
* Instructions on how to use the Mira device
* Urine hCG pregnancy test (at the site of diagnosis) with the Mira kit
* Serum CG pregnancy test (at a UCHealth lab)
* Pregnancy disposition if indicated

Cases:

The follow-up study visits will occur daily for 7 days and include:

* Urine hCG pregnancy test (at home) with the Mira kit. The device will record time of collection.
* Serum CG pregnancy test (at a UCHealth lab)
* Pregnancy disposition

Controls

The follow-up study visits will occur on days 4 and 6 of the menstrual cycle and include:

* Urine hCG pregnancy test (at home) with the Mira kit. The device will record time of collection.
* Serum CG pregnancy test (at a UCHealth lab)
* Pregnancy disposition if identified to be pregnant

B. Description, Risks and Justification of Procedures and Data Collection Tools:

There is the risk that quantitative urine beta hCG testing will not be as sensitive as serum testing. Thus, patients are adequately being monitored according to current standard of care.

Systematic processes and measures that will be employed to minimize patient risks include ensuring patient privacy and protection of Protected Health Information (PHI). Study participants will be thoroughly informed of any possible risks and can decline study participation or to withdraw from the study at any time per standard IRB procedures.

The study team will maintain all research records electronically (REDCap) or in a locked filing cabinet in a secure office. If consent and source documents need to be transported from the clinic to the team offices in the Academic Office Building, the study team will ensure that the documents are securely transported and will not make additional stops between the two buildings.

All research records that identify the participant will kept private to the extent allowed by law. The investigative team maintains the right to keep, preserve, use, and dispose of the findings of this investigation in accordance with IRB guidelines. Investigational records from this study will be maintained in a confidential manner; participant names will not be associated with any published results. Participant information and study information will be pulled from the participant's chart and compiled separately in the REDCap database.

Blood testing is rarely associated with any adverse effects except for discomfort at the blood draw site.

Data Safety Monitoring Plan

The principal investigator will be responsible for the conduct of this study, overseeing participant safety, executing the data and safety monitoring (DSM) plan, and complying with all reporting requirements to local and federal authorities. This oversight will be accomplished through additional oversight from the Data and Safety Monitoring Committee (DSMC) at the University of Colorado Hospital. A summary of the DSMC's relevant activities is as follows:

• Conduct of internal audits Study audits conducted by the DSMC will consist of a review of the regulatory documents, consent forms, and source data verification. Documentation of the audit conducted by the DSMC will then need to be submitted to the IRB of record at the time of the IRB's continuing review of this trial (if applicable per IRB guidelines).

C. Data Analysis Plan: Data will be abstracted and stored on the secure REDCap server at the University of Colorado. Data will be exported into statistical software for descriptive statistics and analyses.

Aim Data source Aim 1: Assess the accuracy and precision of an at-home quantitative urine hCG test in the management of PUL Abstracted hCG measures, timing of measures will be abstracted from both the Mira device and the EPIC EMR Aim 2: Assess patient satisfaction with the Mira at-home quantitative urine hCG test in the management of PUL REDCap survey

Descriptive statistics:

Participant demographic past medical history, gynecologic and obstetric history, as well as study outcomes (urine and serum beta hCG) will be compared between cases and control groups using Pearson Chi-square or Fisher's exact test for categorical factors and present n, percent as summaries. Two-sample t-tests or rank sum tests will be used for continuous measures, as appropriate, and reported as mean and standard deviation or median and interquartile range, respectively. Beta hCG values will be evaluated for distributional assumptions using histograms and Q-Q plot and values will be transformed if necessary to meet assumptions for linear modeling.

Aim1: Assess the accuracy and precision of an at-home quantitative urine b-hCG test in the management of PUL

Comparisons of interest:

1. In controls: evaluate percentage of measurements below the limit of detection, compare between urine and serum beta hCG measurements. Accuracy will be summarized, and McNemar's test will be used to examine agreement between the 2 assays (above vs below limit of detection).
2. In cases: The difference between urine and serum beta hCG values taken on the same day will be the primary outcome of analysis. A linear mixed effects model will be used to evaluate differences in values over the 7 days of measurement (accuracy) and whether the variability if measures over time is constant (precision). Bland-Altman plots will be used to assess not only bias but also the variability across the range of observed values.

Aim2: Assess patient satisfaction with the Mira at-home quantitative urine b-hCG test in the management of PUL.

Descriptive statistics, similar to those described above, will be used to summarize patient satisfaction responses.

D. Summarize Knowledge to be Gained: Findings from this study may have the potential to identify a convenient and accurate method for women to test quantitative urine hCG testing for PUL at home. The findings of this study have a potentially profound impact on the management of PUL and the care and safety of women with this diagnosis.

F. Future Directions: This study will provide pilot data for a future prospective study to assess the sensitivity, specificity, and safety of the Mira home urine pregnancy test in the management of patients with ectopic pregnancy requiring methotrexate for medical management. If the data supports the need for a larger prospective trial, the study team will work closely with campus research leadership to determine the need for an IDE application.

ELIGIBILITY:
Inclusion Criteria for controls:

* Non-pregnant

Inclusion Criteria for cases:

* Diagnosed with PUL requiring ongoing surveillance of serum hCG levels

Exclusion Criteria for controls:

* History of renal disease
* History of type I or type II diabetes
* Known malignancy of any diagnosis including hCG-secreting tumors (hepatobiliary tumors and neuroendocrine tumors) and ovarian germ cell tumors.
* Gestational Trophoblastic Disease
* Use of hormonal contraception within last 3 months
* Patients who work the night shift

Exclusion Criteria for cases:

* History of renal disease
* History of type I or type II diabetes
* Known malignancy of any diagnosis including hCG-secreting tumors (hepatobiliary tumors and neuroendocrine tumors) and ovarian germ cell tumors.
* Gestational Trophoblastic Disease
* Unstable patient, concern for ruptured ectopic pregnancy
* Initial serum hCG level > 100,000 mIU/ml

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 35 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-03-02 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Urine b-hCG | 7 days
  Cases will begin performing urine and serum hCG testing 24 hours after the initial hCG level. Urine hCG testing will be performed on the first morning urine at home and participants will limit water for at least 8 hours before testing. Serum hCG testing will occur at a UCHealth laboratory before 10 am and within 2 hours of the urine test to allow for the comparison of the values. Both urine and serum hCG testing will then occur daily x 7 days, or until a medical or surgical intervention is indicated. If serum testing is indicated on a weekend, patients will present to the UCH Infusion Center.
  Non-pregnant controls will test the first morning urine at home and undergo serum hCG testing in a UCHealth lab on the 4th and 6th day of the menstrual cycle. All urine hCG values will be recorded in the Mira home kit and evaluated in comparison to serum hCG levels.
Serum b-hCG | 7 days
  Cases will begin performing urine and serum hCG testing 24 hours after the initial hCG level. Urine hCG testing will be performed on the first morning urine at home and participants will limit water for at least 8 hours before testing. Serum hCG testing will occur at a UCHealth laboratory before 10 am and within 2 hours of the urine test to allow for the comparison of the values. Both urine and serum hCG testing will then occur daily x 7 days, or until a medical or surgical intervention is indicated. If serum testing is indicated on a weekend, patients will present to the UCH Infusion Center.
  Non-pregnant controls will test the first morning urine at home and undergo serum hCG testing in a UCHealth lab on the 4th and 6th day of the menstrual cycle. All urine hCG values will be recorded in the Mira home kit and evaluated in comparison to serum hCG levels.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
The data of groups after analysis will be shared. We do not need to share individual participant data.